CLINICAL TRIAL: NCT03097666
Title: Clinical Trial to Evaluate Safety and Dose Response Using the C2 CryoBalloon™ Swipe Ablation System for the Treatment of Barrett's Esophagus
Brief Title: Evaluation of Safety and Dose Response Using C2 CryoBalloon™ Swipe Ablation System for Barrett's Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pentax Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0018
Record Dates: First submitted 2017-03-01; First posted 2017-03-31 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Intervention Model Description: Patients with previously untreated (by means of ablation therapy) flat type Barrett's Esophagus (BE) (extent BE ≤C3) with Low-Grade Dysplasia (LGD) or High-Grade Dysplasia (HGD), or residual BE after removal of early adenocarcinoma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- C2 Cryoballoon Swipe Ablation System (Other): C2 Cryoballoon Swipe Ablation System
  Interventions: Device: C2 CRYOBALLOON SWIPE ABLATION SYSTEM

INTERVENTIONS:
Device: C2 CRYOBALLOON SWIPE ABLATION SYSTEM — The C2 CryoBalloon Swipe Ablation System ("CryoBalloon Swipe") is a cryosurgical device with a nitrous oxide cooled balloon probe that is compatible with upper gastrointestinal diagnostic endoscopes.

SUMMARY:
The primary objective is to determine the safety and efficacy of the C2 CryoBalloon™ Swipe Ablation System ("CryoBalloon Swipe") used at increasing doses.

DETAILED DESCRIPTION:
The procedure will be performed on an outpatient basis, and the CryoBalloon Swipe will be used for all ablations following the instructions for use provided with the product.

Patients who meet the eligibility criteria will be assigned to one of the treatment groups and doses, depending on the order of their enrollment:

In phase I, the first 6 patients will be treated with Dose 1 (lowest).

All patients will have to undergo 8 week (±1 week) follow-up EGD to evaluate efficacy of the dose before the study continues.

If the follow-up endoscopies show that Dose 1 eradicates ≥80% of the treated BE (by median percentage) and no SAE's are reported, this dose is defined as the therapeutic dose and enrollment will proceed to phase II.

If Dose 1 eradicates <80% of the treated BE, enrollment in Phase I will continue at the next highest dose. Treatment doses will be escalated in this manner until the earlier of a dose-related Serious Adverse Event (SAE) or determination of the therapeutic dose based on endoscopic exam.

When the therapeutic dose is determined, the study will proceed to Phase II to generate additional safety and efficacy data.

Phase II

Phase II will confirm the safety and efficacy of the therapeutic dose found in Phase I.

---------------------------------------------------------------

Dose-related SAEs include pain in the treatment area greater than 6 (on VAS) on 24 hours and seven (7) days post-treatment; symptomatic stricture requiring an additional EGD with endoscopic dilation before the first follow-up EGD; symptomatic stricture at follow-up EGD; or any stricture (symptomatic or asymptomatic) preventing passage of the diagnostic endoscope at follow-up EGD. Any other serious adverse events within 30 days after treatment will also be evaluated by the Data and Safety Monitoring Board (DSMB) for relationship to the dose and severity.

When a Dose-related serious adverse event occurs, the Holding Rule will be invoked and enrollment at that dose will be held until the DSMB has evaluated the event.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with flat-type (Paris type 0-IIb) BE esophagus, with an indication for ablation therapy, meaning:

   * Diagnosis of LGD or HGD in BE (confirmed by baseline histopathological analysis), OR
   * Residual BE with any grade of dysplasia after endoscopic resection
2. Prague Classification Score C≤3
3. Patients should be ablative-naïve (no previous ablation therapy of the esophagus)
4. Older than 18 years of age at time of consent
5. Operable per institution's standards
6. Provides written informed consent on the IRB-approved informed consent form
7. Willing and able to comply with follow-up requirements

Exclusion Criteria:

1. Esophageal stenosis or stricture preventing advancement of a therapeutic endoscope.
2. Any endoscopically visualized lesion such as ulcers, masses or nodules.
3. History of locally advanced (>T1a) esophageal cancer
4. History of esophageal varices
5. Prior distal esophagectomy
6. Active esophagitis LA grade B or higher
7. Severe medical comorbidities precluding endoscopy
8. Uncontrolled coagulopathy
9. Pregnant or planning to become pregnant during period of study
10. Patient refuses or is unable to provide written informed consent
11. Participation in another study with investigational drug within the 30 days preceding or during the present study
12. General poor health, multiple co-morbidities placing the patient at risk or otherwise unsuitable for trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Dose-related SAEs | 30 days
  Safety will be evaluated by the incidence of Dose-related SAEs. Dose-related SAEs include pain in the treatment area, or any stricture (symptomatic or asymptomatic) preventing passage of the diagnostic endoscope at follow-up EGD.
Efficacy: Percent Eradication by therapeutic dose | 8 weeks
  Eradication percentage of BE confirmed by histological evidence of eradication of BE, after treatment with the therapeutic dose.

SECONDARY OUTCOMES:
Incidence of AEs | up to 30 days post-treatment
  Incidence of all serious and non-serious adverse events up to 30 days post-treatment.
Post-procedure pain | 24 hours and 7 days post-procedure
  Post-procedure pain in the area of the cryoablation treatment (scored on a 0 to 10 point VAS)
Efficacy: Percent Regression | 8 weeks
  Regression percentage at the first follow-up endoscopy, after 1 treatment with the therapeutic dose.
Efficacy: Treatment | 8 weeks
  Efficacy of treatment with CryoBalloon Swipe ablation system, defined as the proportion of patients with ≥80% regression of BE after 1 treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - AMC Medical Research B.V., Amsterdam
  - St. Antonius Hospital Nieuwegein, Amsterdam
  - Catharina Ziekenhuis te Eindhoven, Eindhoven

IPD SHARING:
Plan to Share IPD: No
Data will not be shared.

REFERENCES:
- [Derived] Sunakawa H, Yoda Y, Nonaka S, Suzuki H, Abe S, Ishiguro Y, Ikeno T, Wakabayashi M, Sato A, Nakajo K, Kadota T, Yano T. Prospective multicenter trial of the cryoballoon ablation system for superficial esophageal squamous cell carcinoma on post-endoscopic resection scars: a CRYO-SCAR study (EPOC1902). Gastrointest Endosc. 2024 Sep;100(3):429-437. doi: 10.1016/j.gie.2024.02.018. Epub 2024 Feb 29. PMID 38431103